CLINICAL TRIAL: NCT03377894
Title: Comparison Between Blunt Versus Sharp Expansion of Uterine Incision at Lower Segment Cesarean Section as Regards the Intra-operative Blood Loss & Postoperative Pain
Brief Title: Sharp Versus Blunt Uterine Incision Expansion
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 336695
Record Dates: First submitted 2017-12-10; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group (A) blunt incision (Active Comparator): 100 primigravidas at term who underwent elective transverse lower segment Cesarean section for the first time among the age group of 20 - 37 years with a singleton pregnancy.
  undergoing blunt uterine incision expansion
  Interventions: Procedure: blunt uterine incision expansion
- • Group (B) sharp incision (Active Comparator): 100 primigravidas, at term who underwent elective transverse lower segment Cesarean section for the first time among the age group of 20 - 37 years with a singleton pregnancy undergoing sharp uterine incision expansion
  Interventions: Procedure: sharp uterine incision expansion

INTERVENTIONS:
Procedure: blunt uterine incision expansion — blunt uterine incision expansion
  Arms: • Group (A) blunt incision
Procedure: sharp uterine incision expansion — sharp uterine incision expansion
  Arms: • Group (B) sharp incision

SUMMARY:
comparison between blunt versus sharp expansion of uterine incision at lower segment cesarean section in primigravida as regards the intra-operative blood loss & postoperative pain

DETAILED DESCRIPTION:
the study includes 200 pregnant women, primigravidas, at term who underwent elective transverse lower segment Cesarean section for the first time among the age group of 20 - 37 years with a singleton pregnancy.

The patients are divided randomly into two groups as follows:

* Group (A): undergoing blunt uterine incision expansion
* Group (B): undergoing sharp uterine incision expansion

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy.

Exclusion Criteria:

* previous PID
* any medical or psychiatric
* patients with BMI ≥ 40
* multigravidas
* chronic analgesia use,
* allergy to analgesics,
* multiple pregnancies are also excluded

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
post operative pain | one hour after cs
  Post-operative pain is analyzed by using 4 point verbal rating scale (VRS) which consists of a list of adjectives describing different levels of pain intensity i.e (no pain =1, mild pain = 2, moderate pain = 3, severe pain = 4)
intraoperative bleeding | from skin incision till skin closure
  The intra-operative blood loss is evaluated by towels as follows:
  The surgical towels will be weighed (gm) before and after the operation, and the difference in weight between dry and soaked towels will be calculated. Blood loss during the operation will be calculated by adding the volume of the contents of the suction bottle (ml) to the difference in weight of towels (gm) (weight of soaked towels - weight of dry towels).
The operative time is recorded in minutes | from skin incision till skin closure
  The operative time is recorded in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt